





#### NOTE D'INFORMATION

Etude randomisée de phase III comparant l'association du nivolumab et de l'ipilimumab versus un doublet à base de carboplatine dans le traitement de première ligne du CBNPC avancé chez des patients PS 2 ou de plus de 70 ans eNERGY

N° EudraCT: 2017-002842-60

### Investigateur coordonnateur / principal

Nom: Docteur Hervé Lena

Adresse : Service de Pneumologie - CHU de Rennes - Hôpital de Pontchaillou - 2, rue Henri le Guilloux - 35033

Rennes Cedex 9

Téléphone: 02.99.28.37.38

#### **Promoteur**

Nom: CHU de Rennes

Adresse: Hôpital de Pontchaillou – 2, rue Henri le Guilloux – 35033 Rennes Cedex 9

Principal contact : Direction de la Recherche

Téléphone: 02.99.28.25.55

#### Madame, Monsieur,

Votre médecin vous propose de participer à une étude clinique dont le CHU de Rennes est le promoteur. Avant de prendre une décision, il est important que vous lisiez attentivement ces pages qui vous apporteront les informations nécessaires concernant les différents aspects de cette étude. N'hésitez pas à poser toutes les questions que vous jugerez utiles à votre médecin.

Votre participation est entièrement volontaire. Si vous ne désirez pas prendre part à cette étude, vous continuerez à bénéficier de la meilleure prise en charge médicale possible, conformément aux connaissances actuelles.

#### Pourquoi cette recherche?

Le but de cette étude est de comparer l'efficacité du nivolumab plus l'ipilimumab (aussi appelé Opdivo et Yervoy respectivement) chez des patients atteints de cancer du poumon non à petites cellules métastasique par rapport à une chimiothérapie standard.

Le nivolumab est un nouveau médicament qui bénéficie d'une d'autorisation de mise sur le marché dans le traitement des patients adultes atteints d'un cancer bronchique non-à-petites cellules (CBNPC) localement avancé ou métastatique après une chimiothérapie antérieure.

L'ipilimumab bénéficie quant à lui d'une autorisation de mise sur le marché dans le traitement des patients adultes atteints d'un mélanome avancé (non résécable ou métastatique).

Ces deux molécules sont desanticorps (une protéine humaine) qui peuvent activer le système immunitaire pour l'aider à lutter contre les cellules cancéreuses.

A travers cette étude, nous souhaitons savoir si l'association du nivolumab et de l'ipilimumab est plus efficace que les chimiothérapies recommandées dans votre cas. L'étude concernera des patients atteints d'un cancer du poumon non à petites cellules âgé de plus de 70 ans ou chez qui la maladie entraine une dégradation de l'état de santé.

Nous comparerons également, chez les patients atteints d'un cancer du poumon à un stade avancé, le retard de progression du cancer obtenu avec l'association du nivolumab et de l'ipilimumab et avec les traitements de référence (chimiothérapies).

Nous chercherons également à déterminer si la présence d'une protéine appelée PD-L1 à la surface des cellules cancéreuses des biopsies réalisées pour porter le diagnostic de cancer permet de prédire l'efficacité de l'association du nivolumab et de l'ipilimumab.

Nous vous proposons de participer à cet essai clinique car vous présentez le type de maladie qui pourrait être traité par le protocole que nous proposons dans cette étude.

### Nombre de patients prévu / durée de votre participation

Cette étude est multicentrique, 242 patients participeront à l'essai traités dans plusieurs centres français.

Votre participation est conditionnée par des critères précis d'inclusion et de non-inclusion qui devront être confirmés avant de débuter l'étude.

La durée totale de votre participation sera variable selon la façon dont vous répondrez aux traitements de l'étude. Si vous vous sentez bien avec ces traitements, il est possible que vous participiez jusqu'à 12 mois (1 an) ou plus.

Après l'arrêt de tous les traitements de l'étude (prématuré ou non), il vous sera demandé de revenir pour des visites de suivi afin de surveiller et d'évaluer les effets indésirables ou les éventuels bénéfices qui pourraient être observés suite aux traitements de l'étude (comme il l'est décrit ci-dessous dans la rubrique « suivi », il pourra être nécessaire de recueillir des informations supplémentaires, afin de mieux évaluer la tolérance et l'efficacité des traitements).

#### Traitements étudiés

Cette étude est « ouverte », ce qui signifie que vous saurez quel(s) produit(s) vous recevrez. Au cours de cette étude, vous recevrez :

- ► soit le nivolumab plus l'ipilimumab (Bras « A »),
- ▶ soit une chimiothérapie choisie par le médecin investigateur (Bras « B »).

La chimiothérapie choisie par le médecin investigateur correspond à un traitement de référence pour le cancer du poumon non à petites cellules, composée d'un ou deux produits de chimiothérapie sélectionnés par le médecin investigateur.

Les traitements des bras A et B sont administrés par perfusion intraveineuse (IV), ce qui signifie que le produit est administré par l'insertion d'une aiguille dans une veine de votre bras. Une pompe permettra d'administrer la bonne dose tout au long du temps imparti pour la perfusion.

Si vous remplissez tous les critères requis pour recevoir les traitements de l'étude, vous serez randomisé(e) (c'est-à-dire que l'on vous assignera au hasard) soit dans le bras A (traitement avec nivolumab plus l'ipilimumab), soit dans le bras B (chimiothérapie sélectionnée par le médecin investigateur). Vous avez une probabilité d'une chance sur deux de recevoir le nivolumab plus l'ipilimumab, (en d'autres termes, 1 patient sur 2 sera traité dans le bras A et 1 patient sur 2 sera traité dans le bras B).

Si vous êtes assigné(e) au bras A, vous recevrez le nivolumab à la dose de 240 mg sur 30 minutes et de l'ipilimumab à la dose de 1 mg/kg sur 30 minutes. Le jour de la première administration des deux produits sera appelé « Jour 1 du Cycle 1 ». Selon la réponse de votre organisme au médicament, vous pourrez ensuite recevoir le nivolumab, environ toutes les 2 semaines et l'ipilimumab toutes les 6 semaines. Chaque perfusion durera environ 30 minutes.

Si vous êtes assigné(e) au bras B, vous recevrez la chimiothérapie qui aura été sélectionnée par le médecin investigateur. Ce traitement sera administré par cycle de 3 ou 4 semaines, avec un nombre maximum autorisé de 4 cycles. Le jour de la première administration de chimiothérapie sera appelé « Jour 1 du Cycle 1 » (il y aura donc 3 ou 4 semaines entre « jour 1 du cycle 1 » et « jour 1 du cycle 2 »). Les protocoles de chimiothérapie pourront comprendre :

paclitaxel (90 mg/m2) avec carboplatine (AUC 6) avec une dose qui sera limitée à 700 mg, pendant 4 à 6 heures au Jour 1 de chaque cycle, puis paclitaxel (90/mg/m²) au Jour 8 et au Jour 15 de chaque cycle de 4 semaines,

OU pemetrexed (500mg/m2) avec carboplatine (AUC 5) avec une dose qui sera limitée à 700 mg, pendant 4 à 6 heures au Jour 1 de chaque cycle de 3 semaines,

Si votre maladie répond favorablement après 4 cycles de pemetrexed + carboplatine, le médecin-investigateur pourra vous proposer de poursuivre le pemetrexed seul, en cycles de 3 semaines, sans limite de durée tant que la maladie est contrôlée et que vous supportez bien ce traitement.

## Déroulement de l'étude

Cette étude se déroule en trois grandes phases :

La phase de sélection, pendant laquelle le médecin-investigateur fera des examens afin de déterminer si vous présentez les critères requis pour recevoir les produits de l'étude.

La phase de traitement, pendant laquelle vous recevrez les traitements de l'étude et durant laquelle l'évolution de votre maladie ainsi que les effets indésirables seront observés.

La phase de suivi, débutant après l'arrêt définitif des traitements de l'étude, et qui consiste en des visites de suivi (éventuellement sous forme de contacts téléphoniques) pour surveiller les effets indésirables ou les bénéfices potentiels que vous pourriez avoir avec les traitements de l'étude. Cette phase commencera lorsque le médecin-investigateur estimera que vous n'avez plus de bénéfice à continuer les traitements ou sur votre demande. Elle se terminera soit à votre demande, soit lorsque l'étude sera clôturée.

#### PHASE DE SELECTION

La période de sélection de l'étude dure 28 jours au maximum et peut nécessiter plusieurs visites.

Une fois que le médecin-investigateur aura répondu à toutes vos questions, que vous aurez compris le déroulement de cette étude ainsi que ce document, il vous sera demandé de lire, dater et signer ce formulaire de consentement avant toute procédure liée à l'étude.

Le médecin-investigateur vérifiera que vous pouvez participer à l'étude en examinant vos antécédents médicaux, en vous interrogeant sur les symptômes de votre maladie, en réalisant une consultation complète (examen médical comprenant la mesure des signes vitaux, votre pression artérielle, votre respiration, votre fréquence cardiaque, votre température, votre taille et votre poids). Une détermination de la quantité d'oxygène dans votre sang sera réalisée grâce à un oxymètre de pouls placé au bout d'un doigt (cet examen n'est ni invasif ni douloureux). Le médecin-investigateur vous demandera quels médicaments vous prenez actuellement et avez pris dans le passé, y compris les médicaments vendus sans ordonnance et les herbes médicinales.

Une prise de sang sera faite (20 ml environ) pour réaliser des analyses de routine :

- La numération formule sanguine, appelée aussi hémogramme, qui consiste à mesurer la quantité de globules blancs, de globules rouges et de plaquettes,
- L'analyse de la composition biochimique du sang, appelée aussi Biochimie, qui consiste à mesurer le taux de nombreuses substances chimiques présentes dans le sang, afin de vérifier le bon fonctionnement de votre organisme (reins, foie, glande thyroïde...).
- Egalement, cette prise de sang servira à faire un dépistage de l'hépatite B, C, du VIH et du cytomégalovirus (CMV). Vous ne devez pas avoir été infecté(e) par le VIH et les résultats aux tests des hépatites B et C doivent s'avérer négatifs pour pouvoir participer à cette étude.

Un électrocardiogramme sera réalisé afin d'analyser l'activité de votre cœur.

Un scanner ou une IRM (imagerie par résonnance magnétique) des zones connues de la maladie sera réalisé(e). Ces méthodes radiologiques créent des images de l'intérieur de votre corps qui permettront au médecin investigateur d'évaluer la maladie avant, durant et après les traitements de chimiothérapie ou avec le nivolumab plus l'ipilimumab, et d'observer si la taille des tumeurs varie.

Un scanner ou une IRM du cerveau sera réalisé(e).

Une scintigraphie osseuse sera à réaliser si le médecin investigateur le juge nécessaire. C'est un examen durant lequel une très petite quantité de matériel radioactif est injectée dans une veine de votre bras. Ce matériel est alors transporté par le sang à l'intérieur de vos os et permet de déterminer si le cancer a atteint les os.

Pour les patients âgés de 70 ans et plus à l'entrée dans l'étude, une évaluation gériatrique succincte basée sur des questionnaires usuels sera réalisée.

Si vous pouvez participer à cette étude et que vous le souhaitez toujours, vous reviendrez pour une nouvelle visite avec le médecin-investigateur de l'étude pour entrer dans la phase de traitement.

## PHASE DE TRAITEMENT

Si l'ensemble des résultats des analyses et des procédures effectuées lors la période de sélection vous permet de participer à l'étude, vous reviendrez donc à l'hôpital et les traitements de l'étude vous sera alors assigné :

Si vous êtes assigné(e) au bras A, vous aurez une perfusion intraveineuse de nivolumab, qui durera 30 minutes, suivie d'une perfusion d'ipilimumab qui durera également 30 minutes, la perfusion de nivolumab sera renouvelée toutes les 2 semaines et celle d'ipilimumab toutes les 6 semaines. Les administrations d'immunothérapie auront lieu sous forme de cycles de 6 semaines.

Si vous êtes assigné(e) au bras B, le médecin investigateur vous administrera la chimiothérapie qu'il aura présélectionnée, avec des prétraitements (pour prévenir par exemple les nausées, les vomissements ou les réactions allergiques) en accord avec les pratiques standards. Notez que si vous recevez du pemetrexed, le médecin investigateur vous administrera aussi de l'acide folique et de la vitamine B12 pour limiter la diminution des cellules sanguines et les effets indésirables sur le système gastro-intestinal. Les administrations de chimiothérapies auront lieu sous forme de cycles de 3 ou 4 semaines (jusqu'à 4 cycles), selon le choix de la chimiothérapie.

Si vous ressentez des changements dans votre corps, l'apparition, le développement ou l'aggravation d'un ou plusieurs effets indésirables durant la perfusion, vous devez immédiatement informer le médecin, l'infirmier(e) et un membre du personnel s'occupant de vous.

<u>Durant la période de traitement</u>, avant chaque administration des traitements de l'étude, on vous interrogera sur les signes et les symptômes de la maladie que vous ressentez et les analyses et procédures décrites ci-dessous seront réalisées :

- si, et jusqu'à quel point, la maladie affecte vos activités quotidiennes ;
- quels médicaments vous avez pris ou prenez actuellement, y compris les suppléments à base de plantes et les médicaments sans ordonnance ;

- quels effets indésirables vous avez ressentis. Vous devez signaler à chaque visite à l'hôpital toute apparition et développement, ou aggravation, d'un problème médical (depuis votre dernière visite) au médecin investigateur ou à un autre membre de l'équipe qui s'occupe de vous ;
- un examen physique dont la mesure de votre poids (à chaque visite);
- une mesure des signes vitaux (pression artérielle, fréquence cardiaque, respiration) et une détermination de la quantité d'oxygène dans votre sang seront réalisées à chaque visite demandant une perfusion. Si vous développez une réaction pendant la perfusion, les signes vitaux continueront à être mesurés pour votre sécurité jusqu'à ce que le médecin de l'étude détermine que ce n'est plus nécessaire ;
- un test de grossesse (urinaire ou sanguin) pour les femmes en âge de procréer (les résultats doivent être négatifs pour pouvoir recevoir les produits de l'étude). Après la 1<sup>ère</sup> administration, des tests de grossesse (urinaires ou sanguins) seront réalisés toutes les 6 semaines.
- des prélèvements sanguins (environ 13 ml) auront aussi lieu pour évaluer vos fonctions rénale et hépatique, nombres de globules rouges, de globules blancs et de plaquettes, et pour mesurer votre fonction thyroïdienne (uniquement pour les patients sous nivolumab plus ipilimumab) avant la perfusion des traitements ;
- Votre maladie sera évaluée par scanner ou IRM du thorax, de l'abdomen et du bassin, et si le médecin investigateur le juge nécessaire, un scanner ou une IRM du cerveau et/ou une scintigraphie osseuse seront réalisés. Ces examens seront réalisés toutes les 6 semaines.

En fonction de votre réponse aux traitements et des effets indésirables que vous ressentez, le médecin investigateur pourra vous faire arrêter les traitements de l'étude. Il pourra vous proposer un autre traitement s'il juge qu'il est plus adapté à votre cas.

Dans certains cas, le médecin-investigateur pourra vous proposer de poursuivre l'association nivolumab plus ipilimumab même si la maladie progresse – si ce cas de figure se présente pour vous, le médecin investigateur prendra le temps d'en discuter avec vous et vous remettra une nouvelle fiche d'information et consentement. Vous pouvez aussi, après discussion avec le médecin investigateur, décider d'arrêter les traitements pour d'autres raisons, dont celle de ne plus vouloir être traité(e).

L'arrêt de l'étude pourra être également décidé par le promoteur en cas d'informations nouvelles sur l'efficacité des traitements testés. Votre médecin vous proposera alors un autre traitement adapté à votre situation. Cet arrêt n'aura pas de conséquence sur votre prise en charge par l'équipe médicale.

### PHASE DE SUIVI POST-TRAITEMENT

Visites de suivi initiales n°1 et n°2

Patients traités avec l'association nivolumab plus ipilimumab

Après l'arrêt du nivolumab plus ipilimumab (bras A), vous viendrez à l'hôpital pour les 2 premières visites de suivi. La première visite aura lieu environ 1 mois après l'arrêt des traitements et la seconde approximativement 2 mois plus tard. Durant cette période, le médecin investigateur continuera d'évaluer votre état de santé. Il est important de savoir, par exemple, si vous vous rétablissez ou si vous développez une maladie, ou encore si vous ressentez des effets indésirables. On vous posera les mêmes questions sur votre santé que celles durant votre période de traitement. De même, les procédures (scanners par exemple) et les prélèvements d'échantillons (analyses de laboratoires par exemple) réalisés lorsque vous étiez sous traitement, pourraient être répétés à l'une et l'autre de ces visites de suivi.

Patients traités par chimiothérapie dans l'étude

Si vous avez été traité(e) dans le bras B, avez arrêté tous les traitements anti cancéreux, vous entrerez dans la phase de suivi post-chimiothérapie. Vous viendrez alors à l'hôpital pour les 2 premières visites de suivi. La première visite aura lieu environ 1 mois après l'arrêt des traitements et la seconde approximativement 2 mois plus tard. Durant cette période, le médecin investigateur continuera d'évaluer votre état de santé. Il est important de savoir, par exemple, si vous vous rétablissez ou si vous développez une maladie, ou encore si vous ressentez des effets indésirables. On vous posera les mêmes questions sur votre santé que celles durant votre période de traitement. De même, les procédures (scanners par exemple) et les prélèvements d'échantillons (analyses de laboratoires par exemple) réalisés lorsque vous étiez sous traitement, pourraient être répétés à l'une et l'autre de ces visites de suivi.

#### Visites de suivi supplémentaires (après la visite de suivi n°2)

Ce suivi pourra être effectué à l'occasion de visites avec le médecin investigateur ou par téléphone, tous les 3 mois environ. On vous posera les mêmes questions sur votre santé que lorsque vous étiez sous traitement (nivolumab plus ipilimumab pour les patients du bras A ou chimiothérapie pour les patients du bras B). Pendant cette période, le médecin investigateur continuera d'évaluer votre état de santé. Il est important de connaitre, par exemple, si vous avez récupéré, avez développé une maladie ou ressentez des événements indésirables. Il peut être nécessaire de retourner à

l'hôpital voir le médecin investigateur pour la réalisation de scanners ou d'imagerie supplémentaires comme lorsque vous étiez sous traitement.

Dans le cas où il faudrait évaluer davantage la sécurité d'emploi ou l'efficacité du produit, il peut s'avérer nécessaire d'avoir accès à plus d'informations sur votre état de santé. Le médecin investigateur pourrait tenter d'obtenir ces informations auprès de vous ou de votre médecin traitant. Cela pourra le conduire à vous contacter par courrier ou téléphone.

Dans le cas où le médecin investigateur a besoin d'informations dans le cadre du suivi de l'étude et ne parvient pas à vous joindre, il pourrait être amené à s'enquérir de votre nouvelle adresse, nouveau numéro de téléphone ou des informations sur votre état de santé auprès d'une personne de confiance de votre choix. Si cette personne de confiance n'est-elle même pas joignable, elle peut demander assistance à une tierce personne habilitée à donner uniquement au médecin investigateur des informations limitées à votre patient (nom, dernière adresse connue).

## Ce que l'on vous demandera.

Il est essentiel de respecter vos dates de visite et les instructions du médecin-investigateur et de son équipe.

Si vous participez à cette étude, on vous demandera aussi de bien vouloir :

- décrire votre ressenti et de discuter des éventuels effets indésirables et de tout changement dans votre état de santé;
- informer le médecin investigateur de toute prise de médicaments pendant votre participation à l'étude, qu'ils soient délivrés sur ordonnance ou non (comme des compléments à base de plantes ou des médicaments en vente libre);
- discuter avec lui de tout traitement (avec ordonnance ou en vente libre) que vous souhaiteriez commencer à prendre (avant d'avoir commencé à le prendre) ; certains médicaments ne doivent pas être pris pendant que vous recevez les traitements de l'étude (risque d'interaction provoquant une inefficacité et/ou des effets indésirables). Le médecin investigateur de l'étude vous expliquera quels sont ces traitements. Si vous avez besoin de prendre un de ces médicaments au cours de votre participation à l'étude, vous devez l'informer lui ou le personnel de l'étude. Vous recevrez tous les traitements nécessaires pour votre santé, mais il pourrait être nécessaire d'arrêter les traitements de l'étude si besoin. Ceci est pour votre sécurité.
- annoncer à l'avance au médecin investigateur de l'étude tout traitement médical que vous programmez recevoir pendant l'étude (tel qu'une opération de chirurgie non urgente, par exemple) ;
- annoncer au médecin investigateur de l'étude ou à un membre de son équipe tout changement d'adresse, de numéro de téléphone ou autre information permettant de vous contacter ;

Vous ne pouvez pas participer simultanément à une autre recherche impliquant la personne humaine dans laquelle vous seriez amené(e) à prendre un traitement expérimental tant que vous n'aurez pas arrêté définitivement le produit de l'étude. Vous pourrez participer à une autre recherche impliquant la personne humaine lorsque vous serez en phase de suivi, après une période d'exclusion liée aux nouveaux traitements et déterminée par le médecin-investigateur.

Durant l'étude, vous pourrez éventuellement participer à une autre recherche impliquant la personne humaine sans traitement expérimental sous réserve d'accord préalable du promoteur de l'étude.

#### Risques / Possibles effets indésirables

Les traitements contre le cancer ont souvent des effets indésirables. Certains d'entre eux peuvent être sévères voire mettre en jeu votre pronostic vital. D'autres peuvent encore être inconnus.

Si vous présentez des effets indésirables graves, le médecin-investigateur pourra vous prescrire des médicaments pour traiter ces effets, ou encore retarder les traitements de l'étude ou même l'arrêter définitivement.

Tout nouveau résultat significatif issu de la recherche et survenant au cours de l'étude et qui pourrait influer votre décision de continuer à participer à l'étude vous sera fourni.

## <u>Nivolumab</u>

Le nivolumab peut causer la survenue d'un ou de plusieurs des effets indésirables décrits ci-dessous. Ces informations proviennent de patients atteints de cancer et traités avec le nivolumab dans d'autres essais cliniques. D'autres effets indésirables, non encore connus à ce jour, peuvent également survenir.

Si vous présentez un effet indésirable potentiel, vous devez immédiatement informer le médecin investigateur ou le personnel de l'étude :

| Effets indésirables fréquents | Effets indésirables moins fréquents | Effets indésirables rares mais potentiellement |
|---|---|---|
| | | sérieux |
| | T 0 | |
| Fatigue | Inflammation des intestins | Faible niveau d'oxygène dans le sang |
| Réactions cutanées incluant éruption | Anomalies de la fonction hépatique | Affection ou insuffisance pulmonaire aigue |
| passagère, démangeaisons, urticaire, | (décelées par examens sanguins) | Présence de fluide autour des poumons |
| rougeurs, sécheresse de la peau | Dépigmentation (changement de la | Inflammation de l'appendice (appendicite) |
| Diarrhée | coloration de la peau) | Augmentation des protéines de l'inflammation |
| Nausée | Sécheresse buccale | dans le sang (ex : lipase) |
| Douleurs abdominales | Vomissements | Anomalie des glandes surrénales |
| Perte d'appétit | Perte de poids | Inflammation de l'hypophyse |
| Diminution du nombre de globules | Anomalies de la thyroïde | Modification de l'acuité visuelle (incluant |
| rouges | Anomalies de la chimie sanguine, | baisse ou trouble de la vision), inflammation |
| Fièvre | | oculaire ou saignement dans l'œil |
| Douleurs ou raideurs articulaires | magnésium et du potassium dans le sang | Inflammation du foie |
| | Niveau élevé d'acide urique dans le sang | Affection ou Insuffisance rénale aigue |
| | | Production anormale de globules rouges |
| | voir détails ci- dessous) | Inflammation de la bouche et des muqueuses |
| | | digestives |
| | Vertiges | Gonflement du visage, des bras ou des jambes |
| | Maux de tête | Inflammation du pancréas |
| | Diminution des globules blancs | Mal de dos |
| | | Maladies auto-immunes, incluant le syndrome de |
| | Douleurs, faiblesses, raideurs, spasmes ou | |
| | paralysie musculaires | faiblesse ou paralysie musculaire) |
| | Douleurs dans les bras ou dans les jambes | |
| | Fourmillements, brûlures, | Palpitations cardiaques |
| | engourdissement dans les mains et dans | Inflammation du cœur ou de sa paroi interne |
| | les pieds | Présence de fluide autour du cœur |
| | Essoufflement | Augmentation de la glycémie |
| | Goût anormal | Déshydratation |
| | Rougeurs | Infections : y compris septicémie, infection |
| | | pulmonaire et de la peau |
| | Réaction allergique durant ou entre les | Diminution de la motilité intestinale |
| | <b>F</b> | Désorientation |
| | | Gonflement de la papille optique |
| | aux rayons du soleil | Inflammation du nerf optique |
| | Constipation | Inflammation ou altération de la membrane du |
| | | cerveau et de la moelle épinière |
| | | Réaction au traitement avec rougeurs, anomalies |
| | | des cellules sanguines, augmentation de la taille |
| | augmenter le risque de saignements) | des nodules lymphatiques, et étendue à d'autres |
| | | organes (comprenant le foie, les reins, les |
| | | poumons): |
| | | « syndrome d'hypersensibilité médicamenteuse » |
| | | (DRESS) |

### Inflammation des poumons (pneumopathie)

Il est possible que nivolumab puisse provoquer une inflammation des tissus des poumons. Cet évènement indésirable a été rarement reporté chez des patients traités par nivolumab. Bien que de nombreux patients montrant des anomalies par radiographie ou par scanner n'aient pas eu de symptômes, certains d'entre eux ont développé des symptômes légers à graves, et dans de très rares cas, sont décédés des suites de leur inflammation pulmonaire. Les signes et les symptômes d'une inflammation pulmonaire peuvent inclure : difficulté à respirer, douleur ou inconfort lors de la respiration, douleurs thoraciques, toux, essoufflement, augmentation du rythme respiratoire, fièvre, faible taux d'oxygène dans le sang, fatigue.

Le médecin investigateur et infirmièr(e) vérifieront attentivement tout changement dans votre capacité à respirer ainsi que les autres signes ou symptômes qui pourraient indiquer que vous êtes en train de développer ce type d'inflammation. Il vous sera demandé d'effectuer des tests réguliers, y compris des examens physiques, des mesures de votre taux d'oxygène dans le sang à l'aide d'une technique non invasive (ex: oxymètre de pouls), des tests sanguins, des radiographies thoraciques et/ou des scanners.

Vous devez informer IMMÉDIATEMENT le médecin investigateur ou l'infirmier(e) si vous ressentez un des effets indésirables suivants:

- Tout essoufflement nouveau ou accru.
- Toute douleur thoracique nouvelle ou accrue.
- Toute difficulté respiratoire nouvelle ou accrue.
- Toute toux nouvelle ou accrue ou tout changement important dans votre type de toux, par exemple une augmentation ou une apparition de mucus ou de sang lors d'épisode de toux.
- Un changement dans la quantité d'oxygène dont vous avez besoin.
- Toute fièvre, fatigue ou autres symptômes qui se produisent en même temps qu'un changement de votre respiration ou d'autres symptômes pulmonaires.

Si vous commencez à présenter ces symptômes, le médecin investigateur vous demandera de revenir à l'hôpital pour réaliser des tests supplémentaires (pouvant inclure examen physique, mesure de votre taux d'oxygène dans le sang, tests sanguins, radiographies pulmonaires et/ou scanners).

Toute modification des symptômes pulmonaires sera surveillée de très près et le suivi pourra réclamer votre hospitalisation.

Un traitement spécifique pour contrôler une pneumonie peut s'avérer nécessaire. Vous pourrez également être vu(e) par un pneumologue (médecin spécialiste du système pulmonaire).

Un traitement prolongé avec des médicaments qui suppriment l'inflammation, parfois nécessaire pour gérer les effets indésirables du traitement par nivolumab, peut réduire la capacité de votre corps à lutter contre certaines infections (comme les infections opportunistes, par exemple,). Ces infections peuvent demander un traitement par antibiotique ou par antifongique et engager votre pronostic vital.

Les effets indésirables connus des produits des chimiothérapies possibles dans cette étude (carboplatine, pemetrexed et paclitaxel) sont décrits ci-dessous :

### <u>Ipilimumab</u>

L'ipilimumab peut provoquer un ou plusieurs des effets indésirables énumérés ci-dessous. Cette information est basée sur des données provenant d'autres essais cliniques avec l'ipilimumab chez des patients atteints de cancer. En outre, il peut y avoir des effets indésirables qui ne sont pas encore connus qui peuvent se produire. Vous devez informer votre médecin ou votre infirmière immédiatement sur les éventuels effets indésirables que vous ressentez.

| Effets indésirables fréquents (plus de | Effets indésirables peu fréquents (entre | Effets indésirables rares (<2% mais |
|---|---|---|
| 5% de risque) | 2-5% de risque) | potentiellement graves) |
| <ul> <li>Diarrhée</li> <li>Inflammation du côlon</li> <li>Augmentation des enzymes<br/>hépatiques</li> </ul> | <ul><li>Frissons</li><li>Faiblesse</li><li>Douleurs musculaires</li></ul> | <ul> <li>Diminution des hormones de l'hypophyse</li> <li>Réactions allergiques</li> <li>Inflammation du foie</li> </ul> |
| Fatigue Démangeaisons de la peau Fruption cutanée Nausée Fièvre Perte d'appétit Vomissement Colite Douleur abdominale Maux de tête Constipation Anomalies des glandes | Rougeurs de la peau | <ul> <li>Inflammation de l'hypophyse</li> <li>Diminution des globules rouges</li> <li>Dépigmentation localisée de la peau</li> <li>Diminution ou trouble de la vision ou inflammation de l'œil</li> <li>Engourdissement ou picotement</li> <li>Inflammation de la membrane qui entoure la moelle épinière et le cerveau</li> <li>Inflammation des reins</li> <li>Douleurs articulaires</li> </ul> |
| surrénales • Anomalies de l'hypophyse | | |

Environ 1% des patients traités avec ipilimumab sont décédés des suites d'effets indésirables attribués à l'ipilimumab. Des cas d'infections sévères y compris septicémie (infection du sang qui se traduit par un état inflammatoire généralisé) entraînant parfois le décès, ont été reportés.

### Estomac/intestin:

6 à 12% des patients recevant l'ipilimumab ont eu des réactions auto-immunes sévères au niveau de l'estomac/l'intestin.

Les diarrhées dues au traitement par ipilimumab observées chez les patients peuvent être de minimes à très sévères, avec des saignements ou peuvent, dans de très rares cas, menacer le pronostic vital.

Dans certains cas, la diarrhée a été d'abord d'intensité légère, puis est devenue sévère. Environ 1% des patients ont eu une diarrhée ou des complications au niveau de l'estomac et/ou de l'intestin ayant nécessité l'ablation chirurgicale d'une partie de leur intestin ou ayant entrainé le décès. Dans la plupart des autres cas, l'arrêt de l'ipilimumab et/ou la prise de médicaments (corticoïdes, anti-diarrhéiques) a permis de soigner les diarrhées. La constipation ou des ulcères du gros intestin causés par le traitement par ipilimumab ont été rarement reportés (chez moins de 1% des patients). Si vous savez que vous avez des diverticules (replis de la muqueuse du gros intestin) et/ou une diverticulite (inflammation des diverticules), vous devez informer le médecin investigateur afin qu'il évalue s'il est approprié de vous traiter avec l'ipilimumab.

Manifestations cutanées : la plus fréquente est l'éruption cutanée (rash), la plupart du temps de faible intensité (environ 3 % de cas sévères). Certains patients peuvent avoir des démangeaisons, isolées ou associées à des éruptions cutanées.

Moins de 5% des patients ont présenté un vitiligo (décoloration localisée de la peau, pouvant être définitive). Dans de très rares cas, chez moins de 1% des patients, la formation de vésicules et un décollement de la peau (comme après une brûlure grave) peuvent survenir. Cet état est appelé « syndrome de nécro-lyse épidermique toxique » et peut menacer le pronostic vital et être fatal. Veuillez informer le médecin si vous avez déjà été traité par une thérapie qui active votre système immunitaire contre votre cancer et si vous avez présenté une manifestation cutanée sévère ou ayant menacé votre pronostic vital. Le médecin devra évaluer soigneusement si votre participation à un essai clinique avec ipilimumab est une option appropriée.

Dans de très rares cas (moins de 1% des patients), un syndrome appelé DRESS (qui signifie «Réaction médicamenteuse (ou Rash) avec éosinophilie (augmentation d'une certaine catégorie de leucocytes ou globules blancs) et symptômes systémiques») ou encore « Syndrome d'hypersensibilité médicamenteuse » peut se produire. Les symptômes comprennent : des éruptions cutanées, de la fièvre, l'inflammation des organes internes, le gonflement des ganglions lymphatiques et des anomalies de la formule sanguine. Ce syndrome peut menacer le pronostic vital et être fatal

Vous devez informer le médecin investigateur de tout nouveau rash. Une consultation chez un dermatologue et une biopsie de la peau peuvent être envisagées.

Yeux: Dans de rares cas, (moins de 1% des patients), ipilimumab a causé une inflammation dans les différentes parties de l'oeil ou un changement de couleur de la rétine (fine membrane qui tapisse la face interne de l'oeil). Aucun cas d'atteinte permanente de l'oeil n'a été recensé à ce jour, mais ces évènements pourraient gêner votre vision ou même causer une cécité en l'absence de traitement. Si ces manifestations surviennent, vous aurez peut-être besoin d'un traitement pour réduire l'inflammation. Dans de rares cas (moins de 1% des patients), une vision double peut apparaître en raison d'une faiblesse des muscles oculaires. Vous devrez immédiatement informer le médecin investigateur si vous pensez que votre vue a changé ou si vous développez une vision double ou si vous ressentez une douleur à l'oeil pendant votre participation à cette étude.

Glandes endocrines: environ 3 à 6% des patients prenant l'ipilimumab ont développé des troubles des glandes endocrines (une glande est un ensemble de cellules ou un organe qui sécrète une substance) comme l'hypophyse, la thyroïde ou la glande surrénale. Les atteintes endocriniennes graves ont concerné environ 3% des patients. Les symptômes associés à des troubles de l'hypophyse ou de la glande surrénale sont : fatigue, confusion, perte de poids, troubles de l'érection, et maux de tête. La plupart de ces symptômes ont été contrôlés par une thérapie hormonale ou des corticoïdes.

Foie : Environ 8 à 37% des patients ayant reçu ipilimumab ont présenté des atteintes au foie. Environ 7% des patients ont présenté une toxicité hépatique sévère à la suite d'un traitement par ipilimumab, et environ 1% des cas d'intensité légère à modérée, et dans quelques rares cas ayant mis en jeu le pronostic vital. C'est pourquoi cette étude prévoit des prises de sang fréquentes afin de surveiller votre foie. Une inflammation sévère du foie ayant entraîné le décès est survenu chez moins de 1% des patients traités par ipilimumab. La plupart des cas graves ont été traités efficacement en arrêtant l'ipilimumab et en administrant des anti-inflammatoires tels que des corticoïdes. Vous devrez contacter le médecin investigateur si vous présentez des symptômes qui peuvent être associés à un problème de foie tels que fatigue, faiblesse, vomissement, nausée, coloration jaune de l'oeil ou de la peau, ou douleur abdominale. Des prises de sang plus fréquentes et une biopsie du foie peuvent s'avérer nécessaires si vous souffrez d'anomalies hépatiques graves. Atteintes neurologiques : en de très rares cas (moins de 1 % des patients), une neuropathie motrice liée au système immunitaire (inflammation des nerfs qui contrôlent les muscles), comme le syndrome de Guillain-Barré ou la Myasthénie Grave, peut se produire et mettre en jeu le pronostic vital si elle n'est pas traitée de façon adéquate. Vous devrez informer le médecin investigateur si vous ressentez une faiblesse de vos membres avec ou sans engourdissement ou picotements.

#### Autres événements indésirables:

- Les patients prenant l'ipilimumab ont rarement développé des problèmes touchant simultanément plusieurs organes tels que foie, rein, cœur, muscles, vaisseaux sanguins, œsophage et poumons. Une défaillance aigue des organes entraînant la mort et considérée comme liée à la prise d'ipilimumab s'est produite chez environ 1% des patients.
- Moins de 1% des patients traités par ipilimumab ont eu une méningite (inflammation de la membrane entourant la moelle épinière et le cerveau). La méningite entraîne des maux de tête, des nausées et des vomissements, une raideur du cou, une sensibilité des yeux à la lumière.
- Moins de 1% des patients traités par ipilimumab ont eu une néphrite (inflammation des reins). Les cas de méningites et de néphrites peuvent être résolus en général avec un traitement.
- Par ailleurs, des réactions auto-immunes au niveau de tout autre organe, comme les articulations, peuvent être observées. Elles peuvent causer douleur et gonflement. Moins de 1% des patients traités par ipilimumab ont présenté une douleur articulaire. Dans de rares cas (moins de 1%), il a été reporté, à des degrés variables, une faiblesse des muscles volontaires du corps (myasthénie grave).

#### Autres événements d'intérêt :

Rarement, des patients ont développé une radionécrose (la mort des tissus sains causée par la radiothérapie).

Ces cas ont été signalés chez des patients ayant des antécédents d'irradiation cérébrale pour leur mélanome métastatique. On ne sait pas si cela est dû à la radiothérapie seule ou à l'association de la radiothérapie et d'ipilimumab. La radionécrose cérébrale est un effet indésirable « retard » connu induit par la radiothérapie et est l'une des toxicités tardives post irradiation cérébrale les plus fréquentes. Dans une étude récente de l'ipilimumab administré seul chez des patients présentant des métastases cérébrales issues du mélanome, et dont 31 des 72 patients avaient eu une radiothérapie dans le passé, aucune toxicité neurologique sévère liée à l'ipilimumab n'a été observée.

### Nivolumab en association avec ipilimumab

Compte tenu des informations disponibles à ce jour, les effets indésirables connus du nivolumab en association avec l'ipilimumab sont les suivants :

| Effets indésirables très fréquents | Effets indésirables communs | Effets indésirables non communs | Effets indésirables rares (≥ |
|---|---|---|---|
| (>1/10) | (> 1/100 à < 1/10) | (>1/1.000 à <1/100) | 1/10.000 à < 1/1.000) |
| Augmentation des ALAT : résultat de laboratoire associé avec une fonction hépatique anormale Augmentation des ASAT : résultat de laboratoire associé à une anomalie de la fonction hépatique Diarrhée Fatigue Démangeaisons Nausées Rash | Douleur abdominale Diminution de la fonction de la glande surrénale Augmentation de la phosphatase alcaline : résultat de laboratoire associé à des anomalies du foie ou des os Augmentation de l'amylase : résultat de laboratoire associé à une inflammation du pancréas Diminution de l'appétit Frissons Constipation Toux Augmentation de la créatinine : résultat de laboratoire associé à une diminution de la fonction rénale Déshydratation Etourdissements Sécheresse buccale Sécheresse buccale Sécheresse cutanée Fièvre Perte de cheveux Maux de tête Inflammation de la bouche Inflammation de l'hypophyse Réaction liée à la perfusion Douleur ou raideur articulaire | Réaction allergique Bronchite Dysfonctionnement des nerfs crâniens Diabète Complications du diabète entrainant un excès d'acides dans le sang et un coma diabétique Maladie liée au système immunitaire s'attaquant aux organes en bonne santé Vision double Atteinte hépatique induite par un médicament Sécheresse oculaire Erythème polymorphe : réaction inflammatoire de la peau Syndrome de Guillain-Barré, une maladie auto-immune associée à une faiblesse musculaire progressive ou à une paralysie Augmentation de la fréquence cardiaque Rythme cardiaque anormal Pression artérielle élevée Utricaire Augmentation de la glycémie Inflammation du cerveau, pouvant mettre en jeu le pronostic vital ou être mortelle Inflammation de l'œil | Augmentation de la bilirubine (test sanguin de la fonction hépatique) Insuffisance de multiples organes vitaux tels que le cœur, les poumons, le foie, et les reins. Rhabdomyolyse: libération de fibres musculaires dans la circulation sanguine pouvant endommager vos reins Rosacée: état de la peau semblable à de l'acné entrainant une rougeur du visage Un syndrome associant fièvre, activation et fonctionnement anormal des globules blancs (incluant la destruction d'autres cellules sanguines par certains globules blancs), diminution du nombre de cellules sanguines, rash et augmentation de la taille de la rate. Le syndrome de Stevens-Johnson: trouble inflammatoire de la peau et des muqueuses, entrainant la formation de cloques et une desquamation de la peau Nécrolyse épidermique toxique: maladie potentiellement mortelle caractérisée par des cloques et |

Effet rare (moins de 2%) mais potentiellement sérieux : Un syndrome associant fièvre, activation et fonctionnement anormal des globules blancs (incluant la destruction d'autres cellules sanguines par certains globules blancs), diminution du nombre de cellules sanguines, rash et augmentation de la taille de la rate.

# Carboplatine

| Effets indésirables moins courants (≤ 20%) |
|---|
| Diminution des globules blancs (leucopénie et neutropénie) qui peut vous rendre |
| plus sensible aux infections |
| Diarrhée |
| Constipation |
| Plaies, ulcérations ou plaques blanches dans la bouche (muguet) et la gorge. |
| Douleurs, brûlures ou picotements dans les mains ou les pieds |
| Douleurs, démangeaison, rougeurs, inflammation, gonflement ou plaies au point |
| de perfusion |
| Perte des cheveux |
| Douleur |
| Faiblesse |
| Agueusie (perte de sensibilité au goût) |
| Pâleur |
| Fatigue ou faiblesse inhabituelle |
| Evanouissement ; Etourdissement |
| Changement brusque de la vision, y compris la perception des couleurs |
| Anomalies des tests sanguins évaluant la fonction rénale |
| Augmentation des enzymes hépatiques dans le sang |
| Gonflement du visage, des bras, des mains, des pieds, des chevilles ou des |
| membres inférieurs |
| Essoufflement lors des activités quotidiennes ou en position allongée |
| Bourdonnements dans les oreilles, difficulté d'audition |
| Réaction allergique (éruption cutanée, démangeaisons, rougeurs et gonflements |
| cutanés, essoufflement, et faible pression artérielle) |

# Pemetrexed

| Effets indésirables les plus courants (> 20%) | |
|---|---|
| Fatigue | Diminution des globules blancs (leucopénie et neutropénie) qui peut vous rendre |
| Nausée et/ou vomissements | plus aux infections |
| Perte d'appétit | Diminution des globules rouges (anémie) : cela peut entraîner faiblesse et fatigue |
| | Diarrhée |
| | Rougeurs des plaies dans la bouche, la gorge et sur les lèvres |
| | Infections |
| | Engourdissement, picotements et douleurs des mains et des pieds |
| | Eruption cutanée (rash) |
| | Elévation des enzymes hépatiques dans le sang Gonflement des mains, chevilles, |
| | pieds ou bas des jambes sensible |

# **Paclitaxel**

| Effets indésirables les plus courants (> 20%) | Effets indésirables moins courants (≤ 20%) |
|---|---|
| Diminution des globules blancs (leucopénie et neutropénie) qui peut vous | Ralentissement de la fréquence cardiaque Faible |
| rendre plus sensible aux infections | pression artérielle |
| Diminution des globules rouges (anémie) : cela peut entraîner faiblesse et | Elévation des enzymes hépatiques dans le sang |
| fatigue | |
| Diminution des plaquettes (thrombocytopénie) : peut augmenter le risque | |
| d'ecchymoses, de saignements de nez et des gencives | |
| Infections | |
| Engourdissement, picotements et douleurs des mains et des pieds | |
| Douleurs musculaires et des articulations | |
| Nausées et vomissements | |
| Diarrhées | |
| Rougeurs des plaies dans la bouche, la gorge et sur les lèvres | |
| Perte de cheveux | |

Le médecin investigateur pourra vous donner plus d'informations à propos des effets indésirables listés ci-dessus.

# Autres effets indésirables :

Les prises de sang ou l'utilisation d'un cathéter peuvent avoir les effets indésirables suivants : infection, ecchymoses, rougeur, inconfort ou saignement au point de la piqûre.

Des réactions allergiques aux produits de contraste utilisés lors des examens radiologiques, (scanner ou IRM ou scintigraphie osseuse) peuvent survenir chez des patients (cela reste toutefois rare) et se traduire alors par des démangeaisons ou des éruptions. Dans des cas graves, vous pouvez présenter des difficultés à respirer et une baisse dangereuse de votre pression artérielle. Signalez au médecin-investigateur ou au radiologue toute allergie connue aux produits de contraste, à l'iode ou aux crustacés. Lors de ces examens, vous serez exposé(e) à différents niveaux aux radiations

Certains risques ou des effets indésirables peuvent encore être inconnus à ce jour.

Votre état de santé pourrait ne pas s'améliorer ou s'aggraver pendant que vous participez à cette étude.

Certains médicaments peuvent augmenter la sévérité de ces effets indésirables s'ils sont pris pendant l'étude. Demandez conseil au médecin-investigateur avant de prendre un médicament, quel qu'il soit.

# Risques concernant la procréation, le fœtus et les enfants allaités

### Informations générales

Si vous êtes une femme:

Vous ne devez pas être enceinte ou allaiter et vous ne devez pas débuter une grossesse ou un allaitement pendant que vous êtes sous les traitements de l'étude. Dans le cas spécifique où vous recevriez l'association nivolumab plus ipilimumab, les femmes ne doivent pas allaiter pendant le traitement et jusqu'à 18 semaines après la dernière dose de traitement.

Si vous recevez l'association nivolumab plus ipilimumab, vous devez utiliser une méthode de contraception adéquate afin d'éviter une grossesse pendant toute la durée de cette étude et jusqu'à 23 semaines après la dernière prise de nivolumab plus ipilimumab.

Si vous recevez une chimiothérapie, vous devez utiliser une méthode de contraception adéquate afin d'éviter une grossesse pendant toute la durée de cette étude et jusqu'à 30 jours après la dernière prise de chimiothérapie, ou plus après cette dernière prise si tel est exigé par les Résumés des Caractéristiques Produits (RCP) locaux des produits de chimiothérapie que vous aurez reçus, et conseillé par le médecin investigateur.

Si vous êtes un homme sexuellement actif avec une femme en âge de procréer :

Si vous recevez l'association nivolumab plus ipilimumab, vous devez utiliser une méthode de contraception adéquate pour éviter toute grossesse de votre partenaire et ce, pendant le traitement de l'étude et durant les 31 semaines suivant la dernière prise de nivolumab plus ipilimumab.

Si vous recevez une chimiothérapie, vous devez utiliser une méthode de contraception adéquate pour éviter toute grossesse de votre partenaire et ce, pendant le traitement de l'étude et durant les 6 mois après la dernière prise de chimiothérapie choisie par votre médecin investigateur, ou plus après cette dernière prise si tel est exigé par les Résumés des Caractéristiques Produits (RCP) locaux des produits de chimiothérapie que vous aurez reçus, et conseillé par le médecin investigateur.

Vous devrez immédiatement contacter le médecin investigateur si vous changez de méthode de contraception ou si vous débutez un traitement qu'il ne vous aurait pas prescrit (y compris les médicaments en vente libre et les produits à base de plantes).

#### Risques non prévisibles

Il pourrait exister des risques inconnus pour vous, l'enfant que vous portez ou votre bébé, si vous êtes enceinte, si vous débutez une grossesse ou si vous allaitez pendant l'étude.

#### Résultats de toxicologie de la reproduction en laboratoire et chez l'animal

Bien que des études en laboratoire et chez l'animal aient été réalisées pour évaluer les risques potentiels, elles ne permettent pas de prédire tout ce qui peut se produire chez l'Homme. Aucune étude n'a été menée pour déterminer si le nivolumab ou l'ipilimumab endommagent le matériel génétique (molécules d'ADN). Le nivolumab et l'ipilimumab étant des anticorps, ce risque est considéré comme faible.

De même, aucune étude en laboratoire ni sur des animaux n'a été conduite pour déterminer si le nivolumab ou l'ipilimumab pouvaient s'avérer cancérigènes.

Une étude chez les singes a été réalisée pour évaluer les effets de nivolumab et de l'ipilimumab sur la grossesse. Ces résultats préliminaires ont révélé une augmentation des fausses couches en fin de grossesse et des décès de nouveaunés prématurés. Ces résultats suggèrent un risque potentiel chez l'Homme en cas de poursuite d'un traitement avec nivolumab et/ou ipilimumab pendant la grossesse. Ces résultats anormaux (par exemple, fausses couches chez le

singe) ont eu lieu avec des doses 9 fois supérieures à la dose utilisée dans cet essai à savoir 3 mg/kg de nivolumab toutes les 2 semaines.

#### Informations concernant les grossesses chez l'Homme

L'utilisation de nivolumab ou d'ipilimumab chez la femme enceinte n'a pas été formellement étudiée. Un cas de grossesse a été identifié chez la partenaire d'un homme traité par le nivolumab ou l'ipilimumab. La grossesse s'est déroulée normalement et à la naissance, l'enfant était d'un poids légèrement inférieur à la moyenne.

## Observations portant sur des médicaments similaires de la même classe

Il n'existe aucune information sur des médicaments similaires de la même classe qui pourraient être évalués dans le cadre d'autres études cliniques.

## Observations significatives portant sur le(s) médicament(s) comparateur(s)

Considérant leurs mécanismes d'action, les produits de chimiothérapie disponibles pour le choix du médecin investigateur (carboplatine, paclitaxel, et pemetrexed) peuvent causer des dommages aux fœtus lorsqu'ils sont administrés à la femme enceinte.

Il n'existe pas d'étude spécifiquement menée avec ces produits de chimiothérapie chez la femme enceinte. Chez les animaux, des études ont montré que ces produits de chimiothérapie sont toxiques pour les embryons et des anomalies de développement peuvent alors être générées chez le fœtus.

On ne sait pas si les produits carboplatine, paclitaxelet pemetrexed se diffusent dans le lait maternel.

Les femmes en âge de procréer doivent éviter de débuter une grossesse lorsqu'elles sont sous chimiothérapie (bras B) dans cette étude. Egalement, à cause des risques d'effets indésirables sur l'enfant allaité, il est déconseillé d'allaiter pendant une chimiothérapie.

### Utilisation d'une méthode de contraception interdite par l'étude

Le médecin investigateur vous informera des méthodes de contraception interdites et de celles qui sont acceptables pendant votre participation à cette étude.

Toute méthode de contraception utilisée doit être hautement efficace avec un taux d'échec inférieur à 1% par an, et vous devrez informer le médecin investigateur si vous en débutez une nouvelle pendant l'étude.

#### Exigences concernant les test(s) de grossesse durant l'étude

Si vous êtes une femme susceptible d'avoir des enfants, vous ferez un test de grossesse urinaire ou sanguin dans les 24 heures précédant la première administration des traitements de l'étude, puis toutes les 6 semaines.

### Grossesse ou suspicion de grossesse

Si vous débutez une grossesse, si vous pensez être enceinte, si vous avez un retard de règles ou encore si vous observez un changement au niveau de votre cycle menstruel (comme des saignements plus importants pendant les règles ou des saignements entre les cycles), vous devez immédiatement contacter le médecin investigateur.

# Arrêt d'étude

Si vous débutez une grossesse pendant l'étude, les traitements de l'étude seront immédiatement arrêtés, définitivement, et le médecin investigateur vous orientera vers un obstétricien pour le suivi de votre grossesse, à moins qu'après discussions entre le médecin et le promoteur CHU de Rennes, il soit évalué que le bénéfice de continuer la thérapie prévale sur celui de l'arrêter. Vous continuerez à être suivie pour tout effet indésirable ou bénéfices potentiels liés aux traitements, sous réserve que ce suivi est sans danger pour vous et votre enfant à naître. Le médecin investigateur discutera de cela avec vous ainsi que des options de prise en charge supplémentaire de votre maladie.

Le promoteur n'est pas responsable de la prise en charge financière de la grossesse, de l'accouchement et des soins apportés à l'enfant. Néanmoins, comme il est précisé dans le paragraphe « assurance / Indemnisation », le CHU de Rennes a souscrit une assurance en responsabilité civile couvrant les risques et dommages pouvant résulter de cette étude, dans les conditions de droit commun.

#### Déclaration de la grossesse

Si vous débutez une grossesse pendant l'étude, le promoteur sera tenu informé de cette grossesse et suivra son évolution. Vous serez accompagnée par un médecin compétent afin que celui-ci vous conseille.

#### Informations pour les hommes ayant des partenaires susceptibles d'avoir des enfants

La plupart des traitements expérimentaux n'exposent pas les femmes qui débutent une grossesse à des risques alors que leur partenaire participe à une étude. Cependant, il vous est demandé d'informer le médecin investigateur si votre partenaire débute une grossesse pendant votre participation à cette étude.

Il vous sera demandé, à vous et à votre partenaire, de fournir des informations concernant l'évolution de la grossesse. Le promoteur n'est pas responsable de la prise en charge financière de la grossesse, de l'accouchement et des soins apportés à l'enfant. Néanmoins, comme il est précisé dans la section « assurance / Indemnisation », le CHU de Rennes a souscrit une assurance en responsabilité civile couvrant les risques et dommages pouvant résulter de cette étude, dans les conditions de droit commun.

#### Bénéfices

Les différentes options de chimiothérapie offertes au choix du médecin investigateur dans cette étude (carboplatine-pemetrexed, carboplatine-paclitaxel) sont des traitements de référence pour la plupart des patients éligibles à cette étude. Des bénéfices peuvent être attendus de ces agents de chimiothérapie.

On ne sait pas encore si l'association du nivolumab et de l'ipilimumab peut ou non améliorer votre maladie. Les connaissances obtenues durant cette étude pourront faire progresser la recherche et être utiles à d'autres patients dans le futur.

#### Traitements alternatifs

Il existe d'autres traitements par chimiothérapie disponibles pour votre maladie.

Vous pouvez ainsi décider :

- de recevoir les traitements de référence, sans faire d'essai clinique. Ceci signifie recevoir la thérapie standard pour votre cancer, y compris les produits de chimiothérapie qui font partie des options possibles pour le médecin investigateur dans le bras de traitement B de cette étude,
- de participer à un autre essai clinique,
- de ne pas / plus être traité(e),
- de ne recevoir que des traitements palliatifs. Ces traitements ont pour but de réduire la douleur, la fatigue, la perte d'appétit et autres symptômes causés par votre maladie. Ils ne traitent pas la maladie directement mais à la place essaient d'améliorer votre bien-être. Ces soins tentent de vous garder aussi actif et dans cet état de bien-être que possible. Comme exemples de soins palliatifs pour le cancer du poumon non à petites cellules, on peut citer la thérapie par radiation, ou encore les traitements par biphosphonates ou denosumab qui peuvent diminuer la douleur provoquée par la tumeur lorsqu'elle s'est diffusée aux os.

Discutez de toutes les options avec le médecin investigateur avant de décider de votre participation à cette étude.

#### Assurance / Indemnisation

En accord avec la législation en vigueur, le CHU de Rennes a souscrit une assurance couvrant les risques et dommages pouvant résulter de cette étude dans les conditions de droit commun applicables aux recherches impliquant la personne humaine. Le risque encouru par les femmes enceintes est également couvert par le contrat d'assurance. Le fonds de garantie créé par le législateur pourra également vous couvrir, le cas échéant. En cas de dommage survenant pendant votre participation à l'étude, veuillez immédiatement prendre contact avec le médecin investigateur qui se chargera d'initier les démarches nécessaires auprès des organismes habilités. Si vous subissez un dommage lié à l'étude, l'assurance du promoteur vous indemnisera conformément à la législation en vigueur dans la mesure où ce dommage aura été causé par le produit ou par l'application d'une procédure de l'étude.

Selon les dispositions de l'article L1121-11 du Code de la Santé Publique, vous ne bénéficierez pas d'une indemnisation pour votre participation à cette étude.

# Participation volontaire - Droit de se retirer de l'étude partiellement ou totalement

Votre participation à cette étude est entièrement libre et volontaire.

Selon les dispositions de l'article 1121-11 du Code de la Santé Publique, le médecin investigateur s'assurera que vous bénéficiez d'un régime de sécurité sociale.

Si vous décidez de prendre part à cette étude, vous êtes libre d'arrêter les traitements ou de retirer votre consentement, à tout moment, sans obligation d'en donner la raison et sans que cela n'affecte votre prise en charge médicale.

Toute information recueillie avant le retrait de consentement sera conservée et utilisée pour l'analyse de cette étude sauf opposition de votre part.

La section « Déroulement de l'étude » décrit les visites de suivi que vous pourriez réaliser si vous décidez d'arrêter les traitements de l'étude prématurément.

Dans ce cas, le médecin investigateur n'en déduira pas que vous arrêtez l'étude, mais considérera que vous continuerez à participer au suivi post-traitement décrit dans le paragraphe précité.

Si vous ne souhaitez pas participer à cette période de suivi, vous devez en informer le médecin investigateur par écrit et indiquer clairement quelles évaluations vous ne souhaitez pas effectuer.

### Confidentialité, recueil et utilisation des données

#### Recueil et utilisation des données (données codées)

Dans le cadre de l'étude à laquelle le Dr Léna vous propose de participer, un traitement de vos données personnelles va être mis en œuvre pour permettre l'analyse des résultats de la recherche.

A cette fin, les données médicales et personnelles vous concernant nécessaires à l'étude et notamment des données relatives à vos habitudes de vie et comportements ou votre qualité de vie seront collectées par le médecin investigateur.

Ces données seront identifiées par un numéro de code sans votre nom. Seul le médecin investigateur et son équipe pourra faire le lien entre vos données codées, vous et votre dossier médical.

Les données ainsi codées, seront ensuite utilisées pour l'évaluation scientifique de cette étude et sauf opposition de votre part pourront être utilisées pour d'autres études (actuelles ou futures) portant sur le même produit, une condition médicale identique ou similaire ou toute autre étude jugée pertinente.

Vos données codées pourront être consultées par les Autorités de santé (Agences du médicament française, européenne ou des Etats-Unis par exemple) et toute autre personne requise par la loi, pour vérifier la bonne conduite de cette étude.

Les données collectées pourront être utilisées dans des publications. Cependant, elles resteront codées, sans que jamais votre nom n'apparaisse dans un rapport d'étude ou une publication.

# Accès à votre dossier médical

Pendant l'étude, votre dossier médical, mentionnant votre identité, sera utilisé par le médecin investigateur et son équipe de manière habituelle.

En signant ce consentement, vous autorisez un personnel qualifié et autorisé par le promoteur, les personnes ou sociétés agissant pour son compte, partenaires ou les représentants des Autorités de santé françaises ou étrangères, à consulter votre dossier médical, pour vérifier l'exactitude des données codées collectées dans le cadre de cette étude.

Toutes ces personnes étant soumises au secret professionnel, les informations vous concernant resteront confidentielles.

#### Droits d'accès et de rectification de vos données

Conformément aux dispositions de la loi relative à l'informatique, aux fichiers et aux libertés, vous disposez d'un droit d'accès et de rectification des données vous concernant. Vous disposez également d'un droit d'opposition à la transmission des données couvertes par le secret professionnel susceptibles d'être utilisées et d'être traitées dans le cadre de cette étude.

Vous pouvez accéder directement ou par l'intermédiaire d'un médecin de votre choix à l'ensemble de vos données médicales en application des dispositions de l'article L 1111-7 du Code de la Santé Publique. Cependant, certaines des informations vous concernant pourraient n'être disponibles qu'en fin d'étude.

Ces droits s'exercent auprès du médecin investigateur qui vous suit dans le cadre de cette étude. Vous pouvez en discuter avec lui.

#### Suivi des données après arrêt des traitements et /ou de l'étude

Si votre participation à cette étude est terminée, que la décision ait été prise par vous-même ou par le médecin investigateur, les données précédemment recueillies dans le cadre de l'étude continueront à être utilisées pour les besoins de l'étude, sauf opposition de votre part. En signant le consentement vous autorisez le médecin investigateur ou un membre de son équipe à vous contacter pour vous demander de revenir en visite ou de réaliser des examens supplémentaires pour l'évaluation scientifique de l'étude.

Dans le cas où vous vous retirez explicitement de l'étude, aucune donnée supplémentaire ne sera recueillie à l'exception des données de suivi. Les données d'ores et déjà collectées seront conservées afin de préserver l'intégrité de l'étude.

### Revue par le CPP et l'ANSM

Cette étude a été revue par le Comité de Protection des Personnes du Sud-Ouest et Outre-Mer IV (CPP SOOM IV) et l'Agence Nationale de Sécurité du Médicament et des Produits de Santé (ANSM) qui ont respectivement rendu un avis favorable et une autorisation pour la conduite de cette étude.

### Questions / Informations

Si vous avez des questions concernant l'étude ou vos droits, vous pouvez contacter le médecin investigateur.

Si vous êtes admis(e) aux urgences ou devez être hospitalisé(e), merci d'informer le médecin qui vous prend en charge que vous participez à une recherche impliquant la personne humaine.

Vous serez informé(e) de toute information nouvelle disponible en cours d'étude qui pourrait impacter votre décision de continuer à participer à l'étude.

A l'issue de la recherche, vous pourrez si vous le souhaitez être informé(e) par le médecin investigateur des résultats globaux de celle-ci lorsqu'ils seront disponibles. Par ailleurs, conformément à la loi française, une brève description des résultats sera accessible sur le répertoire public des essais cliniques, sur le site internet de l'ANSM et ce, dans l'année suivant la fin de l'étude dans le monde.

Par ailleurs, une description de cette étude sera disponible en anglais sur le site internet <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, comme requis par la loi américaine, ainsi que sur le répertoire public des essais cliniques, sur le site de l'ANSM (<a href="http://ansm.sante.fr/Services/Repertoire-public-des-essais-cliniques-de-medicaments">http://ansm.sante.fr/Services/Repertoire-public-des-essais-cliniques-de-medicaments</a>), comme exigé par la loi Française. Ces sites ne contiennent pas d'information vous concernant et incluront les résultats globaux de cette étude dans l'année suivant la fin de l'étude dans le monde. Vous pouvez consulter ces sites à tout moment.

Votre médecin traitant sera informé de votre participation à l'étude.

La signature du formulaire de consentement est obligatoire en application de la loi sur les Recherches impliquant la personne humaine (Titre 2 du Livre I du Code de la Santé Publique) et n'affecte aucunement vos droits légaux.

Conformément à réglementation en vigueur, le médecin-investigateur conservera les documents de l'étude au minimum 15 ans après la dernière visite du dernier patient.

#### FORMULAIRE DE CONSENTEMENT

Etude randomisée de phase III comparant l'association du nivolumab et de l'ipilimumab versus un doublet de carboplatine dans le traitement de première ligne du CBNPC avancé chez des patients PS 2 ou de plus de 70 ans eNERGY

N° EudraCT: 2017-002842-60

# Investigateur coordonnateur / principal

Nom: Docteur Herve Lena

Adresse : Service de Pneumologie - CHU de Rennes - Hôpital de Pontchaillou - 2, rue Henri le Guilloux - 35033

Rennes Cedex 9

Téléphone: 02.99.28.37.38

#### **Promoteur**

Nom: CHU de Rennes

Adresse: Hôpital de Pontchaillou – 2, rue Henri le Guilloux – 35033 Rennes Cedex 9

Principal contact : Direction de la Recherche

Téléphone : 02.99.28.25.55

| De Mme/Mr | (Nom de naissance, et nom marital, le cas échéant, en majuscules - Prénom du patient) |
|---|---|
| Le Pr/Dr | |
| | (Prénom, Nom en majuscules - Adresse, n° de téléphone du médecin investigateur) |

m'a proposé de participer à une étude clinique dont le CHU de Rennes est le promoteur. Le but de cette étude est de comparer l'efficacité de l'association nivolumab et ipilimumab et d'une chimiothérapie adaptée chez des patients présentant un cancer du poumon non à petites cellules, récurrent ou métastatique.

Le médecin investigateur m'a expliqué en détail les risques liés au produit de l'étude que je pourrai recevoir. J'ai bien noté que je suis libre d'accepter ou de refuser de participer à l'étude et libre d'interrompre ma participation à tout moment sans donner de raisons et sans conséquence sur la suite de mon suivi médical. Tout autre traitement pourra m'être proposé.

En application de la loi relative à l'informatique, aux fichiers et aux libertés j'accepte, en signant ce formulaire, que les données enregistrées lors de cette étude et des données relatives à mes habitudes de vie et comportements, ma qualité de vie et à mes origines ethniques puissent faire l'objet d'un traitement informatisé par le promoteur ou pour son compte, de façon confidentielle.

J'ai bien noté que le droit d'accès, de rectification et d'opposition au traitement des données me concernant s'exerce à tout moment auprès du médecin investigateur qui me suit dans le cadre de cette étude et que ces données pourront m'être communiquées directement ou par l'intermédiaire d'un médecin de mon choix.

J'accepte également que l'accès direct à mon dossier médical soit donné aux personnes autorisées représentant le promoteur ainsi qu'aux autorités nationales et internationales, dans le cadre d'un contrôle qualité et dans le respect des règles de confidentialité.

J'ai bien noté que les données recueillies dans le cadre de l'étude peuvent être transmises à mon médecin généraliste à ma demande.

J'ai compris que les données pourront être utilisées, sauf opposition de ma part, à des fins scientifiques pour d'autres études (actuelles ou futures) portant sur le même produit, une condition médicale identique ou similaire ou toute autre étude jugée pertinente.

Mon consentement ne décharge pas le promoteur et le médecin investigateur de leurs responsabilités et n'affecte aucunement mes droits légaux.

J'ai bien noté, qu'à l'issue de la recherche, je pourrai, si je le souhaite, être informé(e) des résultats globaux de celle-ci par mon médecin investigateur lorsqu'ils seront disponibles.

Je confirme que j'ai bien reçu toutes les informations sur la nécessité d'éviter absolument toute grossesse pendant l'étude.

Je certifie sur l'honneur être affilié(e) à un régime de sécurité sociale ou bénéficiaire d'un tel régime.

J'ai lu et compris la notice d'information. J'ai pu poser toutes les questions qui me semblaient nécessaires, reçu toutes les réponses à mes questions et eu le temps de réflexion suffisant pour prendre ma décision.

J'ai bien noté que je ne pourrai pas participer simultanément à une autre recherche impliquant la personne humaine portant sur un médicament expérimental pendant la phase de traitement. Je pourrai participer à une autre recherche impliquant la personne humaine lorsque je serai en phase de suivi, après une période déterminée par le médecin-investigateur.

Je reçois un exemplaire de cette note d'information et de ce formulaire de consentement signé. J'atteste n'être ni sous tutelle, ni sous curatelle, ni sous sauvegarde de justice.

### J'ACCEPTE LIBREMENT DE PARTICIPER À CETTE ÉTUDE

Ce document doit être signé, en deux exemplaires originaux, le même jour par le patient et le médecin investigateur.

| Patient: | | |
|---|---|---|
| Prénom, Nom de naissance et nom<br>marital, le cas échéant, en<br>majuscules | Date (à compléter par le patient) | Signature |
| Témoin / Tiers (si le patient ne peu | t pas lire / écrire) : | |
| Prénom, Nom en majuscules | Date (à compléter par le<br>témoin/tiers) | Signature |
| Le Témoin / Tiers doit être totaleme | ent indépendant du médecin investigateu | ır et du promoteur. |
| Médecin Investigateur : | | |
| | | _ |
| Prénom Nom en majuscules | Date | Sionature |

Un exemplaire est à conserver par le médecin investigateur, l'autre exemplaire est à conserver par le patient.